CLINICAL TRIAL: NCT00581477
Title: Treatment of Hypotensive Patients Having a Unique Pattern of Autonomic Symptoms
Brief Title: Treatment of Orthostatic Hypotension
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: 1. enrollment slower than anticipated; 2. FDA approval of droxidopa so no longer need to treat patients on research basis; 3. personnel who were primarily responsible for the study are no longer at Vanderbilt.
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Emily M. Garland, Research Associate Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030750; P01HL056693 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2007-12-27 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Autonomic Nervous System Diseases; Orthostatic Hypotension; Dopamine Beta-Hydroxylase Deficiency; Orthostatic Intolerance
Keywords: autonomic nervous system diseases; blood pressure; congenital; orthostasis; catecholamines
MeSH Terms: conditions — Autonomic Nervous System Diseases; Hypotension, Orthostatic; dopamine beta hydroxylase deficiency; Orthostatic Intolerance; Dizziness | interventions — Droxidopa

STUDY DESIGN:
Intervention Model Description: Although the study was designed as a potential trial of multiple medications, plus placebo, in actuality it served as a means of safely determining the optimal dose of Droxidopa for our patients with Dopamine beta-Hydroxylase Deficiency to take at home. Before each dose of Droxidopa, blood pressure and heart rate were measured for 30 minutes. At 60 or 120 minutes after dosing, blood pressure was also measured after 5 minutes of lying down and 5 minutes of sitting or standing. These measurements were used to calculate the orthostatic change in systolic blood pressure, the primary outcome.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Droxidopa (Experimental): Patients with known or suspected Dopamine beta-Hydroxylase Deficiency were administered Droxidopa doses of 25 mg, 50 mg, 100 mg, 200 mg, 250 mg or 300 mg up to three times daily. Supine and upright blood pressures were subsequently measured 60 to 240 minutes post-dose.
  Interventions: Drug: Droxidopa Oral Product

INTERVENTIONS:
Drug: Droxidopa Oral Product — Droxidopa administered in increasing dosages up to 300 mg
  Other Names: L-DOPS

SUMMARY:
The purpose of this study is to try different medications in patients with low blood pressure and other problems with their involuntary (autonomic) nervous system. The pharmacological trials in this study will perhaps lead to more effective treatment. The protocol includes single dose trials, dose-selection trials, 5-day trials and chronic (approximately 2 months) trials, although only dose-selection trials were consistently performed and have results presented.

DETAILED DESCRIPTION:
We see many patients at the Autonomic Dysfunction Center who can be given a fairly definitive diagnosis, e.g., Orthostatic Intolerance, Pure Autonomic Failure, Multiple System Atrophy, and Baroreflex Failure. However, some patients present with a unique constellation of symptoms of autonomic dysfunction so that they do not fit into a diagnostic category. We hypothesize that a genetic cause exists in some of these patients. We further propose that our comprehensive evaluation of these patients will provide us with information on the pathophysiology of their condition and assist us in optimizing their treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe orthostatic hypotension and other autonomic symptoms who do not meet criteria for one of our standard diagnoses
* non-smokers
* drug-free
* able to give informed consent
* free of pulmonary, renal, hematopoietic, hepatic and cardiac disease

Exclusion Criteria:

* medications affecting the autonomic nervous system
* any chronic illness (cardiac, pulmonary, endocrine, gastrointestinal, rheumatologic)
* anemia (Hct < 30)
* women of childbearing age who are pregnant or nursing
* smokers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Robertson, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight patients with known or suspected dopamine beta-hydroxylase (DBH) deficiency were invited or referred for enrollment in this study.
Pre-assignment Details: Although all 8 patients received droxidopa while in the study, data is not included for 2 patients who had previously been treated with this medication.
Groups:
- Patients With Dopamine Beta-Hydroxylase Deficiency: Patients with known or suspected dopamine beta-hydroxylase deficiency were treated with droxidopa up to 300 mg three time daily. Supine and upright blood pressures were subsequently measured and the length of time the patients were able to stand was ascertained.
Period: Overall Study
Arm/Group | Patients With Dopamine Beta-Hydroxylase Deficiency
Started (Enrolled) | 8 (8 patients were enrolled)
Dose Selection Trial With Droxidopa | 6 (2 patients had been treated with droxidopa prior to enrollment and their data is not included. Since droxidopa restores the norepinephrine that is absent in untreated patients with DBH deficiency, we present only the results for naive patients.)
Droxidopa 25 mg | 6 (Because dosing was individualized for the participants, only 5 of the 6 patients were administered 25 mg of Droxidopa.)
Droxidopa 50 mg | 6 (Because dosing was individualized for the participants, only 5 of the 6 patients were administered 50 mg of Droxidopa.)
Droxidopa 100 mg | 6 (Because dosing was individualized for the participants, only 4 of the 6 patients were administered 100 mg of Droxidopa.)
Droxidopa 200 mg | 6 (Because dosing was individualized for the participants, only 5 of the 6 patients were administered 200 mg of Droxidopa.)
Droxidopa 250 mg | 6 (Because dosing was individualized for the participants, only 2 of the 6 patients were administered 250 mg of Droxidopa.)
Droxidopa 300 mg | 6 (Because dosing was individualized for the participants, only 1 of the 6 patients was administered 300 mg of Droxidopa.)
Completed | 6
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Dopamine Beta-hydroxylase Deficiency
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] — 6 patients with DBH deficiency who had not been treated with droxidopa prior to study enrollment
  years | 19 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure With Standing
Description: The difference between upright and supine systolic blood pressures (dSBP; upright - supine) was calculated for each patient at 60-240 minutes after each dose of droxidopa. For each post-dose timepoint and study day, the average of up to three blood pressure readings per droxidopa dose was calculated. Dosing is individualized for each patient based upon how well the drug is tolerated and the degree of improvement in orthostatic vital signs and symptoms following drug administration. The dosages administered, as well as the number of timepoints and days, therefore, varied between patients.
Time Frame: Up to 240 minutes post dose on Study Days 1, 2, 3 and 4.
Population: Data is missing for 2 participants who had previously been treated with Droxidopa. In addition, since dosing was individualized for each patient, only those participants with data available at the specified timepoint were analyzed.
Measure: Median (Inter-Quartile Range); unit: millimeters of mercury
Groups:
- Droxidopa 25 mg: Participants received up to 3 doses of Droxidopa 25 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
- Droxidopa 50 mg: Participants received up to 3 doses of Droxidopa 50 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
- Droxidopa 100 mg: Participants received up to 3 doses of Droxidopa 100 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
- Droxidopa 200 mg: Participants received up to 3 doses of Droxidopa 200 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
- Droxidopa 250 mg: Participants received up to 3 doses of Droxidopa 250 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
- Droxidopa 300 mg: Participants received up to 3 doses of Droxidopa 300 mg on Study Day 1, 2, 3 or 4. Individual dosing was dependent on how well the drug was tolerated and the degree of improvement in orthostatic signs and symptoms.
Arm/Group | Droxidopa 25 mg | Droxidopa 50 mg | Droxidopa 100 mg | Droxidopa 200 mg | Droxidopa 250 mg | Droxidopa 300 mg
Number analyzed (Participants) | 5 | 5 | 4 | 5 | 2 | 1
millimeters of mercury
  60 minutes post-dose (Day 1) dSBP: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 1
  60 minutes post-dose (Day 1) dSBP | -47 | -39 |  |  |  | -21
  120 minutes post-dose (Day 1) dSBP: number analyzed (Participants) | 4 | 4 | 1 | 1 | 0 | 0
  120 minutes post-dose (Day 1) dSBP | -39.5 [-47.5 to -33] | -35.5 [-62.2 to -10.2] | -24 | -31 |  |
  180 minutes post-dose (Day 1) dSBP: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  180 minutes post-dose (Day 1) dSBP | -38 | -4 |  |  |  |
  240 minutes post-dose (Day 1) dSBP: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0
  240 minutes post-dose (Day 1) dSBP | -47 | -7 |  |  |  |
  60 minutes post-dose (Day 2) dSBP: number analyzed (Participants) | 0 | 0 | 3 | 0 | 0 | 1
  60 minutes post-dose (Day 2) dSBP |  |  | -48 [-51 to -43] |  |  | -30
  120 minutes post-dose (Day 2) dSBP: number analyzed (Participants) | 0 | 0 | 4 | 0 | 0 | 1
  120 minutes post-dose (Day 2) dSBP |  |  | -43.5 [-65.7 to -18.8] |  |  | -13
  180 minutes post-dose (Day 2) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  240 minutes post-dose (Day 2) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  60 minutes post-dose (Day 3) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 0
  60 minutes post-dose (Day 3) dSBP |  |  |  | -51 [-60 to -21] |  |
  120 minutes post-dose (Day 3) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 4 | 0 | 1
  120 minutes post-dose (Day 3) dSBP |  |  |  | -36.5 [-50.2 to -24.8] |  | -23
  180 minutes post-dose (Day 3) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  240 minutes post-dose (Day 3) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  60 minutes post-dose (Day 4) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 1
  60 minutes post-dose (Day 4) dSBP |  |  |  |  | -32.5 [-33 to -32] | -21
  120 minutes post-dose (Day 4) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 1 | 2 | 0
  120 minutes post-dose (Day 4) dSBP |  |  |  | -19 | -47 [-58 to -36] |
  180 minutes post-dose (Day 4) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  240 minutes post-dose (Day 4) dSBP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients stood for upright blood pressure measurements at 60 - 240 minutes following each dose of droxidopa and were asked about adverse events during this time period. Additionally, since patients were inpatient during the study, they were able to report any adverse events throughout the study.
Description: Adverse event information was self-reported by participants and collected for any untoward or unfavorable medical occurrence temporally associated with participation in the research, whether or not considered related to the participant's participation in the research. All-Cause Mortality was not collected with respect to which dose level the patient was currently taking. Orthostatic hypotension and orthostatic symptoms characteristic of DBH deficiency were not considered adverse event.
Groups:
- Droxidopa 25 mg; Droxidopa 50 mg; Droxidopa 100 mg; Droxidopa 200 mg; Droxidopa 250 mg; Droxidopa 300 mg: Patients with known or suspected Dopamine beta-Hydroxylase Deficiency were treated with up to 3 doses per day.
Arm/Group | Droxidopa 25 mg | Droxidopa 50 mg | Droxidopa 100 mg | Droxidopa 200 mg | Droxidopa 250 mg | Droxidopa 300 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2003-11-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT00581477/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT00581477/ICF_001.pdf